CLINICAL TRIAL: NCT01335009
Title: A Study of the Efficacy and PK/PD Relationship of Monotherapy MORAb-004 in Subjects With Metastatic Melanoma
Brief Title: Efficacy Study of Pharmacokinetic(PK)/Pharmacodynamic(PD) Relationship of Monotherapy MORAb-004 in Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-004-201MEL; 2011-001282-40 (EudraCT Number)
Record Dates: First submitted 2011-03-14; First posted 2011-04-13 (Estimated); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; malignant; metastatic
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — ontuxizumab; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MORAb-004, 2 mg/kg (Experimental): Biologic (monoclonal antibody)
  Interventions: Biological: MORAb-004 (monoclonal antibody)
- MORAb-004, 4 mg/kg (Experimental): Biologic (monoclonal antibody)
  Interventions: Biological: MORAb-004 (monoclonal antibody)

INTERVENTIONS:
Biological: MORAb-004 (monoclonal antibody) — Subjects will receive one cycle of treatment with MORAb-004, administered intravenously, on Days 1, 8, 15, and 22 (4 administrations per cycle). Additional cycles will continue without interruption until disease progression occurs or clinical or symptomatic progression as suggested by an investigator.

SUMMARY:
This is a global, Phase 2, open label, dose selection, proof-of-concept study to assess progression free survival in subjects with metastatic melanoma.

Approximately 80 subjects at 29 sites in the U.S., U.K., Germany and Australia will be randomized into one of two dose groups: 2 mg/kg, 4 mg/kg. Weekly treatment will continue until disease progression.

Subjects must have measurable disease by CT Scan or MRI and must have completed at least one prior round of chemotherapy.

Subjects will be assessed for Efficacy, PK/PD, Overall survival, and Safety (Adverse Events/Adverse Events of Interest, Electrocardiograms (ECG's), clinical labs, physical exams/vital signs, tolerability).

DETAILED DESCRIPTION:
MORAb-004 is a monoclonal antibody directed against endosialin, a cell surface glycoprotein, which is expressed on cells involved in tumor vasculature. Studies have found endosialin to play a key role in tumor growth and neovessel formation in numerous cancer types including melanoma. Preclinical pharmacological studies have shown that MORAb-004 is a potentially useful anti-cancer agent. This clinical trial is being performed to determine the efficacy of MORAb-004 at two dose levels in subjects with metastatic melanoma, as well as to establish serum pharmacokinetics and pharmacodynamics of the antibody.

ELIGIBILITY:
Inclusion Criteria:

* Be surgically sterile or consent to use a medically acceptable method of contraception throughout the study period.
* Histologically confirmed diagnosis of metastatic melanoma
* At least 1 prior systemic treatment for metastatic melanoma with disease progression following treatment
* Measurable disease, as defined by RECIST v1.1, assessed within 4 weeks prior to study entry
* At least 3 week interval between first infusion of test article and most recent prior systemic anticancer therapy. All treatment-associated toxicity must be resolved to less than or equal to Grade 1 before the administration of MORAb-004
* Have a life expectancy of at least 3 months as estimated by the investigator
* Have other significant medical conditions well-controlled and stable, in the opinion of the investigator, for at least 30 days prior to Study Day 1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Have sites of disease amenable to the protocol-specified biopsy (Note: All participants will have protocol-specified biopsy at Screening. The second, on-treatment biopsy will be mandatory in the first 30 randomized participants only. For all other participants, the second biopsy is optional.
* Laboratory tests results prior to Study Day 1 within limits as outlined in protocol

Exclusion Criteria:

* Have received no prior systemic treatment for metastatic melanoma
* Evidence of other active malignancy requiring treatment within the last 5 years (other than basal cell or squamous cell carcinoma of the skin), or active brain metastasis
* Clinically significant heart disease (Congestive heart failure of New York Heart Association [NYHA] Class 3 or 4, angina not well controlled by medication, or myocardial infarction within 6 mos.), or ECGs demonstrating clinically significant arrhythmias
* Have any other serious systemic disease, including active bacterial or fungal infection, or any medical condition requiring cytotoxic therapy or chronic (at least 4 consecutive weeks) systemic corticosteroid use
* Have active viral hepatitis or symptomatic Human immunodeficiency virus (HIV) infection
* Be breast-feeding, pregnant, or likely to become pregnant during the study
* Known allergic reaction to a prior monoclonal antibody therapy
* Previous treatment with MORAb-004
* Brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-05-16 (Actual); Primary Completion 2013-12-02 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (20):
  - Pinnacle Oncology, Scottsdale, Arizona
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of Colorado Cancer Center, Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - The University Of Chicago, Chicago, Illinois
  - Oncology Specialists, SC, Park Ridge, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Atlantic Health, Morristown, New Jersey
  - New York University Cancer Institute, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - St. Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (4):
  - Sydney Cancer Center - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Newcastle Melanoma Unit, Calvery Mater Newcastle, Waratah, New South Wales
  - The Crown Princess Mary Cancer Centre, Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
- Germany (3):
  - Universitatsklinikum Essen, Klinik fur Dermatologie, Essen
  - Universitats-Hautklinik, Mainz
  - Eberhard Karls University Tuebingen, Tübingen
- United Kingdom (2):
  - The Royal Marsden Hospital, London
  - Weston Park Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 29 sites in 4 countries (the United States, Australia, Germany, and the United Kingdom), 20 of which enrolled participants.
Pre-assignment Details: A total of 76 participants were randomized to treatment with MORAb-004 (40 participants in the 2 milligram per kilogram [mg/kg] group and 36 participants in the 4 mg/kg group).
Groups:
- MORAb-004 2 mg/kg: Participants received one cycle of treatment with MORAb-004 2 mg/kg, administered intravenously on Days 1, 8, 15, and 22 of the 28-day cycle (4 administrations per cycle). Participants who completed Cycle 1 continued with additional cycles without interruption or dose escalation until disease progression, using computed tomography/magnetic resonance imaging (CT/MRI) or until they discontinued the study for any reason. Participants were assessed for disease progression by CT/MRI every 8 weeks from the date of first study treatment (that is, Cycle 1 Day 1), regardless of delays in treatment.
- MORAb-004 4 mg/kg: Participants received one cycle of treatment with MORAb-004 4 mg/kg, administered intravenously on Days 1, 8, 15, and 22 of the 28-day cycle (4 administrations per cycle). Participants who completed Cycle 1 continued with additional cycles without interruption or dose escalation until disease progression, using CT/MRI or until they discontinued the study for any reason. Participants were assessed for disease progression by CT/MRI every 8 weeks from the date of first study treatment (that is, Cycle 1 Day 1), regardless of delays in treatment.
Period: Overall Study
Arm/Group | MORAb-004 2 mg/kg | MORAb-004 4 mg/kg
Started | 40 | 36
Completed | 9 | 3
Not Completed | 31 | 33
Not completed — Too ill to travel to study sites | 1 | 0
Not completed — Death | 28 | 32
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least one dose of study medication, analyzed by the actual treatment received.
Groups:
- MORAb-004 2 mg/kg: Participants received one cycle of treatment with MORAb-004 2 mg/kg, administered intravenously on Days 1, 8, 15, and 22 of the 28-day cycle (4 administrations per cycle). Participants who completed Cycle 1 continued with additional cycles without interruption or dose escalation until disease progression, using CT/MRI or until they discontinued the study for any reason. Participants were assessed for disease progression by CT/MRI every 8 weeks from the date of first study treatment (that is, Cycle 1 Day 1), regardless of delays in treatment.
- Total: Total of all reporting groups
Arm/Group | MORAb-004 2 mg/kg | MORAb-004 4 mg/kg | Total
Number analyzed (Participants) | 40 | 36 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (12.22) | 61.2 (12.15) | 63.3 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 27
  Male | 22 | 27 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 39 | 32 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 39 | 34 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival (PFS) at Week 24
Description: PFS was defined as the time (in weeks) from the date of randomization to the date of the first sign of disease progression (PD) based on Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1, or date of death, regardless of cause. PD greater than or equal to (>=) 20 percent (%) increase in the nadir of total tumor burden (TTB) (minimum 5 millimeter [mm]). Participants who were alive with no disease progression had their PFS time censored at the date of their last tumor assessment. Participants who received a new anti-cancer therapy before disease progression had their PFS time censored at the date of their last tumor assessment before the new anti-cancer therapy was started. PFS was analyzed using Kaplan Meier method.
Time Frame: Week 24
Population: Primary efficacy population included all participants in the safety population who meet all key eligibility criteria (including measurable disease at baseline after at least 1 systemic treatment) analyzed by the dose level to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MORAb-004 2 mg/kg | MORAb-004 4 mg/kg
Number analyzed (Participants) | 39 | 36
percentage of participants | 13.5 [5.0 to 26.4] | 8.9 [2.3 to 21.3]

2. Secondary Outcome: Percentage of Participants With PFS at Weeks 16 and 52
Description: PFS was defined as the time (in weeks) from the date of randomization to the date of the first observation of PD (RECIST version 1.1) or date of death, regardless of the cause. PD >=20% increase in the nadir of TTB (minimum 5 mm). Participants who were alive with no disease progression had their PFS time censored at the date of their last tumor assessment. Participants who received new anti-cancer therapy before disease progression had their PFS time censored at the date of their last tumor assessment before the new anti-cancer therapy was initiated. PFS was based on the Kaplan-Meier method.
Time Frame: Week 16 and Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MORAb-004 2 mg/kg | MORAb-004 4 mg/kg
Number analyzed (Participants) | 39 | 36
percentage of participants
  Week 16 | 32.5 [18.3 to 47.6] | 20.8 [9.2 to 35.7]
  Week 52 | NA [NA to NA] — Data from pre-specified Kaplan Meier estimation was inestimable, because of no available participants with events at Week 52. | 8.9 [2.3 to 21.3]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in weeks) from the date of randomization to the date of death, regardless of cause. In the absence of death confirmation, or for participants alive at the time of analysis, the survival time was censored at the date of the last study follow-up. OS was calculated using the Kaplan-Meier method. As per planned analysis, efficacy outcomes was planned to be analyzed until cut-off date (02 December 2013).
Time Frame: Date of first study treatment (Day 1) to date of death or up to approximately 2 years 7 months
Population: Primary efficacy population included all participants in the safety population who meet all key eligibility criteria (including measurable disease at baseline after at least 1 systemic treatment) analyzed by the dose level to which they were randomized. Participants without documentation of death at the time of analysis were censored at the date last known to be alive.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MORAb-004 2 mg/kg | MORAb-004 4 mg/kg
Number analyzed (Participants) | 39 | 36
weeks | 40.9 [29.0 to 53.3] | 29.3 [22.9 to 35.4]

4. Secondary Outcome: Percentage of Participants With Overall Response
Description: ORR was defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) that occurred (defined by RECIST version 1.1) using CT/MRI. Per RECIST 1.1, CR= disappearance of all lesions; PR greater than or equal to (>=) 30percent (%) decrease from baseline in TTB. As per planned analysis, efficacy outcomes was planned to be analyzed until cut-off date (02 December 2013).
Time Frame: Date of first study treatment (Day 1) to complete response or partial response, assessed up to approximately 2 years 7 months
Population: ORR population included a subset of participants from the primary efficacy population who had at least 1 on-study radiologic evaluation performed (in addition to their baseline evaluation), analyzed by the dose level received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MORAb-004 2 mg/kg | MORAb-004 4 mg/kg
Number analyzed (Participants) | 34 | 32
percentage of participants | NA [NA to NA] — Data was inestimable, because of no available participants with events at Week 52. | 3.1 [0.0 to 9.2]

5. Secondary Outcome: Optimal Biologic Dosing (OBD) of Morab-004
Description: OBD is defined as the dose level/exposure level at which three parameters are met: 1) adequate pharmacokinetic (PK) profile with a serum half-life (t1/2) of >=48 hours, 2) at least minimal demonstration of antitumor efficacy (50% or greater PFS rate at 16 weeks), and 3) change of 25% or greater from baseline value in any of the pharmacodynamic (PD) parameters assessed in the study in 30% of participants at that dose level.
Time Frame: Day 1 Cycle 1 (Cycle length = 28 days)
Population: All participants in the safety population who receive at least one dose of MORAb-004 and who had at least one on-treatment PK/PD assessment performed that is sufficient to evaluate the endpoint of interest. Here "overall number of participants analyzed" are participants who were available for this outcome measure.
Measure: Number; unit: milligram(s)
Arm/Group | MORAb-004 2 mg/kg | MORAb-004 4 mg/kg
Number analyzed (Participants) | 39 | 36
milligram(s) | NA — Here 'NA' signifies that OBD was not evaluated due to minimal antitumor efficacy (less than 50%) and percentage of participants with response was too low hence, was not demonstrated. | NA — Here 'NA' signifies that OBD was not evaluated due to minimal antitumor efficacy (less than 50%) and percentage of participants with response was too low hence, was not demonstrated.

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 45 days after the last dose of study drug (up to approximately 8 years 11 months)
Description: Safety population included all randomized participants who received at least 1 dose of study drug, analyzed by the actual treatment received. The severity of AE toxicities was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria, v4.03, where applicable.
Arm/Group | MORAb-004 2 mg/kg | MORAb-004 4 mg/kg
All-Cause Mortality (participants affected / at risk) | 28/40 | 32/36
Serious Adverse Events (participants affected / at risk) | 17/40 | 16/36
Other Adverse Events (participants affected / at risk) | 40/40 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MORAb-004 2 mg/kg (N=40) | MORAb-004 4 mg/kg (N=36)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Tumour haemorrhage (Infections and infestations) | 0 (0) | 1 (1)
Delirium (General disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MORAb-004 2 mg/kg (N=40) | MORAb-004 4 mg/kg (N=36)
Fatigue (General disorders) | 18 (28) | 18 (28)
Chills (General disorders) | 13 (13) | 18 (20)
Pyrexia (General disorders) | 9 (11) | 12 (17)
Infusion related reaction (General disorders) | 4 (4) | 1 (3)
Oedema peripheral (General disorders) | 4 (4) | 3 (6)
Influenza like illness (General disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (18) | 15 (21)
Constipation (Gastrointestinal disorders) | 9 (11) | 9 (9)
Vomiting (Gastrointestinal disorders) | 3 (3) | 9 (12)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 6 (10)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 3 (4)
Headache (Nervous system disorders) | 21 (35) | 21 (31)
Dizziness (Nervous system disorders) | 3 (4) | 4 (4)
Tremor (Nervous system disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 9 (14) | 11 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 8 (16) | 10 (22)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4)
Confusional state (Psychiatric disorders) | 0 (0) | 4 (6)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (3)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Feeling cold (General disorders) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 2 (2)
Localised oedema (General disorders) | 0 (0) | 1 (2)
Pain (General disorders) | 1 (1) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram RR interval prolonged (Investigations) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (2) | 0 (0)
QRS axis abnormal (Investigations) | 1 (1) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 2 (2)
Specific gravity urine increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (10) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (2)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (2) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 2 (4)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Fungating wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 2 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (5)
Atrial flutter (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctival oedema (Eye disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No